CLINICAL TRIAL: NCT04966936
Title: The Effect of Different Microprocessor Knee Prostheses on Mobility and Gait Parameters in Unilateral Traumatic Transfemoral Amputees
Brief Title: The Effect of Different Microprocessor Knee Prostheses on Mobility and Gait Parameters in Transfemoral Amputees
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Physical Medicine and Rehabilitation Specialist, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Other Study IDs: 17
Record Dates: First submitted 2021-07-02; First posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-06

CONDITIONS: Amputation
Keywords: Transfemoral Amputee; microprocessor knee prostheses
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Unilateral traumatic transfemoral amputee patients using C-Leg prosthesis: The activity levels of the patients will be evaluated by the Amputee Mobility Predictor, the mobility of the patients by the Locomotor Capacity Index, the prosthesis satisfaction in general with the visual analog scale (VAS), the walking ability and capacity with the prosthesis will be evaluated by the 2 min walking test, and the gait analysis will be evaluated in the motion analysis laboratory.
  Interventions: Other: questionnaires for clinical assessments; Other: 2 minute walking test; Other: The gait analysis at the motion analysis laboratory.
- Unilateral traumatic transfemoral amputee patients using Genium prosthesis: The activity levels of the patients will be evaluated by the Amputee Mobility Predictor, the mobility of the patients by the Locomotor Capacity Index, the prosthesis satisfaction in general with the visual analog scale (VAS), the walking ability and capacity with the prosthesis will be evaluated by the 2 min walking test, and the gait analysis will be evaluated in the motion analysis laboratory.
  Interventions: Other: questionnaires for clinical assessments; Other: 2 minute walking test; Other: The gait analysis at the motion analysis laboratory.
- Unilateral traumatic transfemoral amputee patients using Genium-X3 prosthesis: The activity levels of the patients will be evaluated by the Amputee Mobility Predictor, the mobility of the patients by the Locomotor Capacity Index, the prosthesis satisfaction in general with the visual analog scale (VAS), the walking ability and capacity with the prosthesis will be evaluated by the 2 min walking test, and the gait analysis will be evaluated in the motion analysis laboratory.
  Interventions: Other: questionnaires for clinical assessments; Other: 2 minute walking test; Other: The gait analysis at the motion analysis laboratory.

INTERVENTIONS:
Other: questionnaires for clinical assessments — Amputee Mobility Predictor, Locomotor Capacity Index, visual analog scale (VAS)
Other: 2 minute walking test — the individual is asked to walk in his natural course within 2 minutes on a track whose distance is measured beforehand, and at the end of two minutes, the distance he walks will be recorded in meters (m).
Other: The gait analysis at the motion analysis laboratory. — Temporo-spatial parameters (gait speed (m/s), cadence (step/s), other foot contact (%), double support time (second), single support time (second), stance phase time (sec), swing phase time (sec), stride length (meters)) and kinematic parameters (hip, knee, ankle joint angles (frontal, sagittal, transverse plane), maximum knee flexion angles in the stance and swing phase, velocity-dependent maximum knee flexion angles in the swing phase, knee flexion moments will be compared

SUMMARY:
Microprocessor knee joints are prosthetic knee joints with an integrated processor or a computer that can analyze data. During walking, parameters such as step speed, joint angles, and weight transferred through sensors are analyzed by the computer inside the joint and determines the movement for the safest and most normal walking. They have different features from each other in terms of weight/height, sensor and processor frequency, load carrying capacity, phase control (hydraulic, pneumatic, magnetic), battery properties, water resistance, and special activity mode. C-Leg, Genium, Genium X3, Rheo Knee 3, Rheo Knee XC, Orion etc. prostheses of different companies are used as oscillating and compression phase microprocessor knee prostheses.

Publications on C-leg, Genium and Genium X3 prostheses are limited in international literature. Although there are existing studies comparing C-leg and Genium, there is no study comparing these three prostheses. The investigators think that our study is important because it is the first study in the literature to compare these three prostheses. In this study, the investigators aimed to examine the effects of different microprocessor knee prostheses on mobility and gait parameters in unilateral traumatic transfemoral amputees.

DETAILED DESCRIPTION:
The study will be carried out with patients who applied to the outpatient clinic or who received inpatient treatment in the orthopedic rehabilitation (amputee) clinic. The patient's demographic information (age, gender, height, weight, body mass index, education level, occupation, marital status) and clinical characteristics (amputation date, cause of injury, amputation side, etc.) will be recorded with the evaluation to be made to the patient. The activity levels of the patients will be evaluated by the Amputee Mobility Predictor, the mobility of the patients by the Locomotor Capacity Index, the prosthesis satisfaction in general with the visual analog scale (VAS), the walking ability and capacity with the prosthesis will be evaluated by the 2 min walking test, and the gait analysis will be evaluated in the motion analysis laboratory.

ELIGIBILITY:
Inclusion Criteria:

1. be over 18 age
2. Having a unilateral traumatic transfemoral amputation for at least 3 months
3. Using prosthesis for at least 3 months
4. Not having cognitive problems
5. Using your current prosthesis for at least 4 hours a day
6. No concomitant orthopedic problem in the contralateral lower extremity

Exclusion Criteria:

1. Under the age of 18
2. Presence of neurological, cardiovascular and pulmonary disease that may affect walking performance
3. Being inadequate in Turkish communication
4. Residual extremity skin loss
5. Using a walking aid

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: 27 unilateral traumatic transfemoral amputee patients (9 patients using C-Leg prostheses, 9 patients using Genium prostheses, 9 patients using Genium-X3 prostheses)
Sampling Method: Non-Probability Sample
Enrollment: 27 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Amputee Mobility Predictor | Through study completion, an average of 1 month
  The amputee is evaluated with 21 functions and a score is obtained. According to this score, the patient's K activity level is determined. K0: The patient is immobile, does not have the potential and ability to ambulate or transfer with the prosthesis. K1: The patient can use the prosthesis for ambulation and transfers. Prostheses provide limited or unlimited in-home ambulation. K2: The patient provides limited ambulation in the community with the prosthesis. K3: The patient has the potential to use the prosthesis at variable speeds. The patient can use the prosthesis not only for ambulation, but also for occupation, therapeutic activities and exercises. K4: The patient has the potential and ability to use the prosthesis in high-energy activities.
Locomotor Capacity Index | Through study completion, an average of 1 month
  the patient's ability to perform 14 activities with the prosthesis is evaluated. The total maximum score is 42, and the higher the total score, the higher the locomotor capacity.
visual analog scale | Through study completion, an average of 1 month
  The visual analog scale is a 10 cm long line and patients are asked to mark a point on this line that they deem appropriate according to the degree of satisfaction (0: not at all satisfied with the prosthesis, 10: the highest satisfaction with the prosthesis)
The 2-minute walk test | Through study completion, an average of 1 month
  In this test, the individual is asked to walk in his natural course within 2 minutes on a track whose distance is measured beforehand, and at the end of two minutes, the distance he walks is recorded in meters (m).
Temporo-spatial parameters of the patients in the motion analysis laboratory | Through study completion, an average of 1 month
  gait speed (m/s), cadence (step/s), other foot contact (%), double support time (second), single support time (second), stance phase time (sec), swing phase time (sec), stride length (meters)
kinematic parameters of the patients in the motion analysis laboratory | Through study completion, an average of 1 month
  hip, knee, ankle joint angles (frontal, sagittal, transverse plane), maximum knee flexion angles in the stance and swing phase, velocity-dependent maximum knee flexion angles in the swing phase, knee flexion moments

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Özcan, MD, Principal Investigator — Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Locations (1):
- Gaziler Physical Medicine and Rehabilitation Education and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No